CLINICAL TRIAL: NCT06415591
Title: Auricular Neuromodulation in Veterans With Fibromyalgia: A Randomized, Sham-Controlled Study
Brief Title: Auricular Neuromodulation in Veterans With Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F5050-R; I01RX005050 (NIH)
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia
Keywords: Pain; Fibromyalgia; Magnetic Resonance Imaging; Veterans; Percutaneous Electrical Nerve Field Stimulation; Vagus Nerve
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either true or sham PENFS using the auricular device (series of 4, weekly placement with ongoing 5 day (M-F) stimulation - manufacturer recommended) treatments, then assessed for changes in pain and function at 12 and 24 weeks post-treatment. The 12-week time point is chosen to evaluate longer-term neural changes as an indicator of neural plasticity, given the continued improvements seen in the investigators' PENFS group based on preliminary data. The 24- week timepoint is chosen to evaluate longer term (6 months) pain outcomes related to PENFS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, sham placebo controlled. Randomization will be performed by a research coordinator, who will assign each participant a study number and keep a record of whether they are receiving true or sham PENFS, thus maintaining blinding of the participant, the study physicians, the research assistant, and the data analysis team including the P.I. (A.W.) until completion of the follow-up period and data analyses can be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- True PENFS (Active Comparator): Percutaneous electrical nerve stimulation applied to the ear x 4 over a 4 week period. The device is placed over the area of the ear and worn home continuously for a 5-day period, during which time it stimulates at a pre-set on/off duty cycle. At each in-person visit, the device is replaced until the device has been placed 4 times. The stimulation delivered is below the threshold of sensory perception.
  Interventions: Device: Percutaneous electrical nerve field stimulation
- Sham PENFS (Sham Comparator): A device is placed at the same points for the same amount of time and at the same intervals as the true device. This device will not deliver electrical stimulation.
  Interventions: Device: Percutaneous electrical nerve field stimulation

INTERVENTIONS:
Device: Percutaneous electrical nerve field stimulation — FDA-approved acupuncture-like therapy applied to the external ear targeting several cranial nerve branches including the auricular branch of the vagus nerve to improve pain, physical function, and reduce symptoms of opioid withdrawal.
  Other Names: PENFS

SUMMARY:
PENFS (percutaneous electrical nerve field stimulation) is an FDA-cleared acupuncture-like therapy applied to the external ear targeting several cranial nerve branches including the auricular branch of the vagus nerve to improve pain, physical function, and reduce symptoms of opioid withdrawal. PENFS has been previously shown to provide improvements in fibromyalgia, a difficult to treat chronic pain syndrome, which correlate with changes observed using a special kind of MRI called resting state functional connectivity MRI (rs-fcMRI) that evaluates brain activity at rest. The goals of this study are to rigorously test the initial promising results of PENFS in a much larger group of Veterans suffering from fibromyalgia and to identify potential mechanisms of PENFS effects. Further developing non-pharmacologic therapies for pain can help to improve quality of life and function for those suffering from fibromyalgia and decrease reliance on opioids and other drugs that have numerous side effects for individuals suffering from chronic pain.

DETAILED DESCRIPTION:
BACKGROUND: In the setting of the opioid epidemic, it is crucial to develop and assess non-pharmacologic treatments for pain and understand underlying mechanisms. In the present investigation, the investigators assess a novel non-pharmacologic approach to chronic pain treatment in Veterans suffering from fibromyalgia (a notoriously difficult to treat pain syndrome that affects 5-10 million Americans and disproportionately affects those returning from the Gulf War), utilizing brain imaging as a biomarker and heart rate variability (HRV) to assess a vagal mechanism. Preliminary results from prior VA-funded feasibility study reveal a trend towards improved pain and function with a FDA-approved, non-pharmacologic therapy - auricular percutaneous electrical nerve field stimulation (PENFS) - over standard therapy control for Veterans suffering from fibromyalgia, correlating to altered network connectivity on rs-fcMRI (resting state functional connectivity MRI). PENFS-related improvements continued through 12 weeks following the completion of treatment and correlated to changes in cross-network connectivity, which differed between groups. Based on the preliminary data, the investigators now intend to rigorously assess the treatment effects of PENFS in a large, double-blind, randomized, sham-controlled study.

OBJECTIVE: The proposed Merit, a randomized, sham-controlled trial of auricular PENFS, evaluates the clinical utility of PENFS for fibromyalgia as compared to sham placebo control, acute and longitudinal PENFS-related neural changes visualized on rs-fcMRI and effects of PENFS on HRV as a potential vagal mechanism of pain relief.

HYPOTHESIS: True PENFS results in non-placebo-related short-and long-term pain and physical function improvements that can be correlated with altered connectivity and HRV.

METHODS: For Aim 1, 240 total participants meeting 2016 diagnostic criteria for fibromyalgia (male and female, age 18-60 years old) will be randomized to either true (n=120) or sham (n=120) auricular PENFS.

Neuroimaging data, self-reported pain, and physical function will be assessed at baseline and at 1- and 12- weeks post-treatment to evaluate neural correlates of PENFS-related treatment. Participants who meet study criteria will be randomized to either true or sham PENFS (series of 4, weekly) treatments and assessed for rsfcMRI and functional changes at 1- and 12-weeks post-treatment. Baseline and follow-up rs-fcMRI will be utilized to identify biomarkers of fibromyalgia and PENFS treatment effects for Aim 2 in a subset of 62 participants from Aim 1 who qualify for MRI procedures. Cardiopulmonary data will be simultaneously collected during rs-fcMRI and utilized for the exploratory Aim 3 to evaluate potential PENFS effects on HRV as an outcome measure for vagal effects. In the initial phase preliminary analytical validation will be accomplished in the first 30 participants following IRB approval, hiring and training of staff, and establishment of an image processing pipeline. If initial milestones are met, the rigorous, double-blind, sham-controlled study in a larger group of Veterans will continue. Veterans who are initially assigned to sham placebo PENFS and are not identified as placebo-responders will be offered the opportunity to test the true PENFS device. This study addresses the critical need to clinically evaluate non-pharmacologic therapies for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older; for those who participate in the MRI portion, age 20-60 years old (limit specifically set for participants receiving an MRI scan; limit set to minimize brain structural changes due to aging)
* For those who participate in the MRI portion, right-handedness, to provide consistency in brain structure and function (limit specifically set for participants receiving an MRI scan; limit set to minimize brain structural changes due to aging)
* For those who participate in the MRI portion, the ability to safely tolerate MRI
* Diagnosis of fibromyalgia by the American College of Rheumatology 2016 criteria69
* Pain score of 4 or greater on DVPRS51 in the 3 months prior to enrollment
* Intact skin in area of PENFS treatment

Exclusion Criteria:

* Pregnancy (self-reported)
* History of seizures or neurologic conditions that alter the brain
* Claustrophobia, MRI-incompatible implants, or other conditions incompatible with MRI (only for those who participate in MRI)
* History of uncontrolled psychiatric illness, autoimmune disease that leads to pain, or skin conditions that can increase risk of infection at PENFS site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Improvements in Clinical Pain (DVPRS) | Through study completion, an average of 1 year
  The investigators will assess whether pain and functional improvements occur with the application of PENFS. Clinical pain, as measured by the Defense Veterans Pain Rating Scale (DVPRS), will be our primary outcome. This measure is rated on a scale of 0 to 10, with 0 being "no pain" and 10 being "as bad as it could be, nothing else matters". Assessments will be administered at baseline, immediately pre- and post-treatment (the device is replaced every 5 days for a total of 4 device applications), 12 weeks post-treatment, and 24 weeks post-treatment.
Improvements in Clinical Pain (Self-reported analgesic consumption) | Through study completion, an average of 1 year
  The investigators will assess whether pain and functional improvements occur with the application of PENFS. Changes in clinical pain will also be assessed for this outcome via self-reported analgesic consumption. This measure is not rated on a scale - it is self-reported use. Assessments will be administered at baseline, immediately pre- and post-treatment (the device is replaced every 5 days for a total of 4 device applications), 12 weeks post-treatment, and 24 weeks post-treatment.

SECONDARY OUTCOMES:
rs-fcMRI as a biomarker of treatment response | Baseline, 12 weeks post-treatment
  Resting state functional connectivity magnetic resonance imaging (rs-fcMRI) will be performed at baseline and 12 weeks post-treatment to assess changes in cross-network connectivity with the default mode network (DMN) and sensorimotor network (SMN) as well as connectivity within the salience network (SN).
PENFS effects on parasympathetic tone as measured by heart rate variability (HRV) | Baseline, 12 weeks post-treatment
  Heart rate variability (HRV) will be assessed at the MRI scans at baseline and 12 weeks post-treatment with an MR-compatible pulse oximeter to evaluate the effects of PENFS on parasympathetic tone.
Changes in Fibromyalgia Severity (FIQ-R) | Through study completion, an average of 1 year
  Fibromyalgia severity will be assessed via the Fibromyalgia Impact Questionnaire (FIQ-R). Each question is rated on a scale of 1 to 10 with 1 being the least impact/severity and 10 being the most impact/severity. Assessments will be administered at baseline, immediate post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
Functional Improvements (Arm curls) | Through study completion, an average of 1 year
  Functional improvements will be assessed using the arm curl test. Assessments will be administered at baseline, immediate post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
Changes in Fibromyalgia Severity (PSD) | Through study completion, an average of 1 year
  Fibromyalgia severity will be assessed via the Polysymptomatic Distress Scale (PSD). This measure ranges from scores of 0 to 31, with 0 being the least severe and 31 being the most severe. Assessments will be administered at baseline, immediate post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
Patient Reported Improvements (PROMIS change) | Through study completion, an average of 1 year
  Patient reported improvements will be assessed using the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) measures. PROMIS measures are rated on a scale of 1 to 5 with 1 being the least intense ("Never") and 5 being the most intense ("Always"). Assessments will be administered at baseline, immediate post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.
Functional Improvements (30-s chair stand) | Through study completion, an average of 1 year
  Functional improvements will be assessed using the 30-s chair stand. Assessments will be administered at baseline, immediate post-treatment, 12 weeks post-treatment, and 24 weeks post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Woodbury, MD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Woodbury PAIN Lab Page — https://www.woodburypainlab.com/